CLINICAL TRIAL: NCT01214694
Title: Rehabilitation Research and Training Center for Traumatic Brain Injury Interventions--Internet-based Interacting Together Everyday, Recovery After Childhood TBI
Brief Title: Internet-based Interacting Together Everyday, Recovery After Childhood TBI (I-InTERACT)--RRTC
Acronym: I-InTERACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: MetroHealth Medical Center (Other); Nationwide Children's Hospital (Other); Rainbow Babies and Children's Hospital (Other); Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: H133B090010--02
Record Dates: First submitted 2010-09-01; First posted 2010-10-05 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Traumatic Brain Injury
Keywords: TBI; intracranial edema; brain edema; craniocerebral trauma; head injury; brain hemorrhage, traumatic; subdural hematoma; brain concussion; head injuries, closed; epidural hematoma; extra-axial hemorrhage; cortical contusion; Additional relevant MeSH terms:; Nervous System Diseases; Wounds and Injuries; Disorders of Environmental Origin; Central Nervous System Diseases; Trauma, Nervous System; Brain Diseases; Brain Injuries
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Edema; Craniocerebral Trauma; Brain Hemorrhage, Traumatic; Hematoma, Subdural; Brain Concussion; Head Injuries, Closed; Hematoma, Epidural, Spinal; Brain Contusion; Nervous System Diseases; Wounds and Injuries; Disorders of Environmental Origin; Central Nervous System Diseases; Trauma, Nervous System; Brain Diseases; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Active Comparator: Internet Resources Comparison (IRC) (Experimental): Participants will receive the Internet resource comparison group treatment
  Interventions: Behavioral: Internet Resources Comparison (IRC)
- I-InTERACT (Experimental): Participants will receive a 24 week, 27 session internet-based parenting skills program
  Interventions: Behavioral: Internet-based Interacting Together Everyday: Recovery After Childhood TBI (I-InTERACT)
- I-InTERACT Express (Experimental): Participants will receive an abbreviated 7 week, 14 session version of the I-InTERACT parenting skills program.
  Interventions: Behavioral: Internet-based-Interacting Together Everyday, Recovery after Childhood TBI Express (I-InTERACT Express)

INTERVENTIONS:
Behavioral: Internet-based Interacting Together Everyday: Recovery After Childhood TBI (I-InTERACT) — Families in I-InTERACT will view 10 web-sessions (like chapters) and participate in 27 family meetings over the course of 24 weeks focusing on increasing positive parenting skills, reducing parenting stress, and improving child behavior problems. Meetings will be conducted in their home using a computer hook-up with a trained therapist.
  Other Names: I-InTERACT
  Arms: I-InTERACT
Behavioral: Internet-based-Interacting Together Everyday, Recovery after Childhood TBI Express (I-InTERACT Express) — Families in I-InTERACT Express will view 10 web-sessions (like chapters) and participate in 14 family meetings over the course of 7 weeks focusing on increasing positive parenting skills, reducing parenting stress, and improving child behavior problems. Meetings will be conducted in their home using a computer hook-up with a trained therapist.
  Other Names: I-InTERACT Express
  Arms: I-InTERACT Express
Behavioral: Internet Resources Comparison (IRC) — Families in the IRC group will receive computers, high speed internet access, and links to brain injury information and resources. The resources are available for families to access as often as they choose.
  Other Names: IRC
  Arms: Active Comparator: Internet Resources Comparison (IRC)

SUMMARY:
The purpose of this study is to test two on-line interventions for families of young children who have experienced moderate or severe traumatic brain injury (TBI). This project builds upon the investigators' previous research by modifying the online intervention content to address the needs of young children with TBI. The goal of this project is to develop an intervention that will encourage positive parenting behaviors, improve child behaviors, and reduce parent distress and burden following TBI. The investigators hypothesize that the intervention groups will exhibit more effective parenting skills as well as better child functioning and lower levels of parental distress at follow-up than will the active comparison group.

DETAILED DESCRIPTION:
The investigators will conduct a multi-site randomized controlled trial (RCT) comparing the efficacy of 7-week Internet-based Interacting Together Everyday, Recovery after Childhood Traumatic Brain Injury Express (I-InTERACT Express) and 24-week long web-based positive parenting skills programs Internet-based Interacting Together Everyday, Recovery after Childhood Traumatic Brain Injury (I-InTERACT) to an internet resource group (IRC) involving access to internet resources and education about brain injury. The project builds upon the feasibility and efficacy findings from an ongoing randomized trial comparing the efficacy of a 24-week positive parenting skills program to access to internet resources. However, it differs in size and scope by including multiple sites, and by including an abbreviated parenting skills training arm in response to family feedback that the existing 24-week intervention was excessively long, resulting in adherence difficulties. The investigators anticipate that the improvements in parenting skills and psychological functioning will translate into improved parent-child relationships and reductions in child behavior problems. Over time, such improvements in child and parent functioning should contribute to academic and social success and more successful community integration.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe TBI that occurred within the last 24 months
* Overnight hospital stay
* English-speaking
* Parent must be willing to provide informed consent

Exclusion Criteria:

* Child does not live with parents or guardian
* Child or parent has history of hospitalization for psychiatric problem
* Child suffered a non-blunt injury (e.g., projectile wound, stroke, drowning, or other form of asphyxiation)
* Diagnosed with moderate or severe mental retardation, autism, or a significant developmental disability

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 117 (Actual)
Dates: Start 2009-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Parent Report Measures | 5 years

SECONDARY OUTCOMES:
Neuropsychological Testing | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Shari L Wade, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; H. Gerry Taylor, PhD, Principal Investigator — Rainbow Babies and Children's Hospital; Keith O. Yeates, PhD, Principal Investigator — Nationwide Children's Hospital; Michael Kirkwood, PhD, Principal Investigator — Children's Hospital Colorado; Terry Stancin, PhD, Principal Investigator — MetroHealth Medical Center
Locations (5):
- United States (5):
  - The Children's Hospital, Denver, Aurora, Colorado
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio

REFERENCES:
- [Derived] Aguilar JM, Cassedy AE, Shultz EL, Kirkwood MW, Stancin T, Yeates KO, Taylor HG, Wade SL. A Comparison of 2 Online Parent Skills Training Interventions for Early Childhood Brain Injury: Improvements in Internalizing and Executive Function Behaviors. J Head Trauma Rehabil. 2019 Mar/Apr;34(2):65-76. doi: 10.1097/HTR.0000000000000443. PMID 30499926
- [Derived] Wade SL, Cassedy AE, Shultz EL, Zang H, Zhang N, Kirkwood MW, Stancin T, Yeates KO, Taylor HG. Randomized Clinical Trial of Online Parent Training for Behavior Problems After Early Brain Injury. J Am Acad Child Adolesc Psychiatry. 2017 Nov;56(11):930-939.e2. doi: 10.1016/j.jaac.2017.09.413. Epub 2017 Sep 14. PMID 29096775